CLINICAL TRIAL: NCT07323680
Title: A Phase 1, Open-Label, 2-Period, 2-Formulation, Within-Subject Crossover Comparative Pharmacokinetic, Pharmacodynamic, and Safety Study of 1 Dose Level of Aspirin for Injection and Oral Aspirin Tablets in Healthy Adult Human Subjects Under Fasting Conditions.
Brief Title: Comparative Pharmacokinetic, Pharmacodynamic, and Safety Study of 1 Dose of Aspirin for Injection and Oral Aspirin Tablets in Healthy Adult Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Rhoshan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Rho-11-003
Record Dates: First submitted 2025-12-18; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Aspirin; DNA modification methylase phi3TII, Bacteriophage phi-3T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rho-11 administered in Period 1, oral aspirin administered in Period 2 (Experimental)
  Interventions: Drug: 325 mg Oral Aspirin; Drug: 325 mg aspirin by rapid IV push
- Oral aspirin administered in Period 1, Rho-11 administered in Period 2 (Experimental)
  Interventions: Drug: 325 mg Oral Aspirin; Drug: 325 mg aspirin by rapid IV push

INTERVENTIONS:
Drug: 325 mg Oral Aspirin — Drug: aspirin 325mg
  • Subjects will be administered 325 mg aspirin orally
Drug: 325 mg aspirin by rapid IV push — Drug: Rho-11 Subjects will be administered 325 mg aspirin by rapid IV push
  Other Names: Rho-11

SUMMARY:
The purpose of this study is to compare the safety, pharmacokinetics, and pharmacodynamic effects of aspirin administered intravenously with aspirin administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must meet all of the following criteria to be enrolled in this study:

  1. Healthy males and non-pregnant and no breast-feeding females, ≥ 18 and ≤ 55 years of age (on the day of Informed Consent).
  2. Non-smokers or past smokers (having ceased smoking at least 6 months before the first dosing).
  3. Body Mass Index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 on the day of screening.
  4. The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at Screening.
  5. The subject has a hemoglobin level with the following acceptable range at Screening: (Male: 12.8 to 17.4 g/dL (128 to 174 g/L); Female: 10.8 to 15.0 g/dL (108 to 150 g/L).
  6. The subject has liver function tests within normal limits or has results that do not show clinically significant abnormalities, as judged by the investigator at Screening.
  7. The subject has estimated glomerular filtration rate eGFR (CKD-EPI) ≥50 mL/min (0.833mL/sec/1.73m2) at Screening.
  8. Acceptance of use of contraceptive measures during the whole study by both female and male subjects.
  9. No tattoo, body piercing or any cosmetic treatment involving skin penetration within 90 days before screening, unless evaluated by Investigator as non-significant for inclusion in the study.
  10. The subject agrees to comply with all protocol requirements.
  11. The subject can provide written informed consent.
  12. The subject must fluently speak and understand Czech.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. The subjects has had any major illness within 3 months before dosing with study drug or any significant ongoing chronic medical illness, as judged by the investigator.
  2. The subjects has a history of active deep vein thrombosis and/or thromboembolic disorder, including history of hypothrombinemia and vitamin K deficiency.
  3. The subject has a history of neuropsychiatric disease, hypertension, cardiac failure, cerebrovascular disease, chronic respiratory disease, asthma, nasal polyps associated with asthma, hepatic or renal impairment, recent dehydration (within last 30 days), gout thyrotoxicosis or systemic lupus erythematosus and other connective tissue disorders.
  4. The subject has a history of gastrointestinal bleeding or has active gastrointestinal disease that could affect drug absorption.
  5. The subject has a history of hemorrhagic disorder.
  6. Prothrombin time or activated partial thromboplastin time level outside the normal range at screening and check-in.
  7. The subject has an increased risk of bleeding including but not limited to: any history of a clinically significant bleeding problem, any recent (within 30 days preceding the first dose of study drug) major trauma, platelet count <100,000 mm3
  8. The subject has a history of glucose-6-phosphate dehydrogenase deficiency.
  9. The subject has a recent history of tooth extraction within 3 weeks before dosing with study drug.
  10. The subject is a smoker or has used nicotine-containing products (e.g., snuff, nicotine patch, nicotine chewing gum, mock cigarettes, inhalers, or "vape" devices) within 6 months before the first dose of study drug and throughout the study (including the washout period).
  11. The subject has a history of alcohol abuse or drug addiction within 1 year prior to check-in or excessive alcohol consumption (regular alcohol intake >21 units per week for male subjects and >14 units of alcohol per week for female subjects), or use of alcohol 48 hours before dosing with study drug.
  12. The subject has a positive test result for drugs of abuse, alcohol, or cotinine at screening or before dosing with study drug.
  13. The subject has used any prescription (excluding hormonal birth control) or over-the-counter medications, including fish oil and other herbal or nutritional supplements and, in particular, aspirin (no aspirin-containing medications allowed at all), nonsteroidal anti-inflammatory agents (No NSAIDS allowed at all, and no acetaminophen, diclofenac, ketorolac allowed), or anticoagulation therapy within 14 days before dosing with study drug and throughout the entire study period (including the washout period).
  14. The subject has received vaccination against Varicella zoster within 6 weeks before dosing with study drug.
  15. The subject has a positive test result for COVID-19, hepatitis B surface antigen, hepatitis C virus antibody, or HIV type 1 or 2 antibodies at screening.
  16. The subject has received the COVID-19 vaccine within 14 days before Day -3, or subjects who plan to receive a COVID-19 vaccine at any time during the study.
  17. The subject has a history of relevant drug and/or food allergies (i.e., allergy to aspirin or any excipients, allergic skin reactions, or any significant food allergy that could preclude a standard diet in the clinical unit).
  18. The subject has consumed grapefruit or grapefruit juice, Seville orange or Seville orange-containing products (e.g. marmalade), or alcohol-, caffeine-, poppy-, or xanthine-containing products within 48 hours.
  19. The subject is involved in strenuous activity or contact sports within 24 hours before dosing with study drug and during the study.
  20. The subject has donated blood or blood products >450 mL within 30 days before dosing with study drug.
  21. The subject has received study drug in another investigational study within 30 days or 5 half-lives, whichever is longer, before dosing with study drug.
  22. In the opinion of the investigator, the subject is not suitable for entry into the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum thromboxane B2 from baseline | 1 hour before dosing and 2, 5, 10, 20, 30, 45, 60, and 180 minutes post dosing]
  Change in serum thromboxane B2 from baseline to 180 minutes post treatment

SECONDARY OUTCOMES:
Urinary 11-dehydro-TXB2 levels | Every 12 hours from 24 hours prior to dosing to 72 hours after dosing.
  Measured levels of 11-dehydro-TXB2 in urine following treatment
Urinary 2,3-dinor-6-keto-PGF1alpha | Every 12 hours from 24 hours prior to dosing to 72 hours after dosing.
  Measured levels of 2,3-dinor-6-keto-PGF1alpha in urine following treatment
Acetylsalicylic Acid Plasma Pharmacokinetics | 1 hour prior to dosing, and 1,3,5,10,15,20,30, and 45 minutes and 1,1.5,2,3,6,8, and 24 hours postdosing.
  Measured change in levels of acetylsalicylic acid in plasma following treatment
Salicylic Acid Plasma Pharmacokinetics | 1 hour prior to dosing, and 1,3,5,10,15,20,30, and 45 minutes and 1,1.5,2,3,6,8, and 24 hours postdosing.
  Measured change in levels of salicylic acid in plasma following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Purvis, MD, Study Director — jpurvis@rhoshanpharma.com
Locations (1):
- Quinta-Analytica s.r.o., Prague, Czechia

IPD SHARING:
Plan to Share IPD: No